CLINICAL TRIAL: NCT04365621
Title: The Clinical and Socio-demographic Characteristics of Young People Aged 12 to 25 Consulting on Ambulatory Structures in the Seine Saint-Denis
Acronym: EPS-12-25
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Januel (Other)
Responsible Party: Sponsor-Investigator, Januel, Psychiatrist, head of the clinical research department, Centre hospitalier de Ville-Evrard, France
Organization: Centre hospitalier de Ville-Evrard, France (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10477M-EPS-12-25-2020
Record Dates: First submitted 2020-04-16; First posted 2020-04-28 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Psychosis
Keywords: psychiatry- mental illness-young population- ultra-high risk of psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: It is a prospective study with a single group assignement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ultra-high risk of psychosis patient (Other): patient with ultra -high risk of psychosis will be enrolled to the study
  Interventions: Other: we enrolled ultra-high risk of psychosis (UHR) patient to describe

INTERVENTIONS:
Other: we enrolled ultra-high risk of psychosis (UHR) patient to describe — there is no intervention because we study only the prevalence of patients meeting UHR criteria

SUMMARY:
A prospective study of the clinical and socio-demographic characteristics of young people aged 12 to 25 consulting on ambulatory structures in the Seine Saint-Denis.

This research project, intersectoral and inter-institutional, built in a territorial logic, is therefore intended to study longitudinally over a year the population of young consultants in the different units participating in it, to highlight their common profiles and differences.

This will be the first clinical research work concerning adolescents and young adults using mental health services in the Seine Saint Denis Ouest.

DETAILED DESCRIPTION:
The main objective of the study will be to quantify the rate of subjects seeking help in our units meeting the criteria of subject with an ultra-high risk of psychosis (UHR).

Secondary objectives:

* Observe the transition rate of these high risk patients at one year.
* Study the socio-demographic and general psychopathology profiles of 12 - 25 year olds using the services of CMP, CASADO, mobile team and RCL.
* Monitor the development of school and professional integration, the overall functioning and self-esteem of subjects at six months and one year.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls consulting in the structures involved in the study of the Seine-Saint-Denis department.
* Aged 12 to 25.
* Patients with an ultra high risk of psychosis.
* Affiliated with social security or with State Medical Aid (AME).

Exclusion Criteria:

* Subject with known neurological pathology
* Subject with insufficient knowledge of French

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 900 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-05-02 (Estimated); Study Completion 2021-05-02 (Estimated)

PRIMARY OUTCOMES:
Rate of ultra-high risk mental | "Month 1"
  Rate of subjects meeting the criteria for subjects with an ultra-high risk mental state after passing the CAARMS to M1.
Rate of ultra-high risk mental | "Month12"
  Rate of subjects meeting the criteria for subjects with an ultra-high risk mental state after passing the CAARMS to M12.

SECONDARY OUTCOMES:
16-Item Version of the Prodromal Questionnaire (PQ-16) | J0
  developed to facilitate screening in subjects consulting in classical clinical practice of the risk of developing psychosis
Rosenberg Scale | "Month 1"
  Chosen because brief (10 items),which can be supplemented by subjects from different age groups and backgrounds, without weighing down the clinical interview with the young subject.
Rosenberg Scale | "Month 6"
  Chosen because brief (10 items),which can be supplemented by subjects from different age groups and backgrounds, without weighing down the clinical interview with the young subject.
Rosenberg Scale | "Month 12"
  Chosen because brief (10 items),which can be supplemented by subjects from different age groups and backgrounds, without weighing down the clinical interview with the young subject.
Adolescent Depression Rating Scale (ADRS) | Day 0
  10-item hetero questionnaire created specifically to assess depression in adolescence. The ADRS has demonstrated good validity and improved ability to discriminate against depressed and not depressed adolescents
Adolescent Depression Rating Scale (ADRS) | Month 6
  10-item hetero questionnaire created specifically to assess depression in adolescence. The ADRS has demonstrated good validity and improved ability to discriminate against depressed and not depressed adolescents
Adolescent Depression Rating Scale (ADRS) | Month 12
  10-item hetero questionnaire created specifically to assess depression in adolescence. The ADRS has demonstrated good validity and improved ability to discriminate against depressed and not depressed adolescents
Social and Occupational Functionning Assessment Scale (SOFAS) | "Day 0"
  cited in the DSM-V to assess the V axis and overall functioning, ranging from 0 to 100 on a continuum ranging from "superior functioning in a large number of activities" to "inability to maintain minimal hygiene, inability to operate without significant outside assistance."
Social and Occupational Functionning Assessment Scale (SOFAS) | "Month 6"
  cited in the DSM-V to assess the V axis and overall functioning, ranging from 0 to 100 on a continuum ranging from "superior functioning in a large number of activities" to "inability to maintain minimal hygiene, inability to operate without significant outside assistance."
Social and Occupational Functionning Assessment Scale (SOFAS) | "Month12"
  cited in the DSM-V to assess the V axis and overall functioning, ranging from 0 to 100 on a continuum ranging from "superior functioning in a large number of activities" to "inability to maintain minimal hygiene, inability to operate without significant outside assistance."
Comprehensive Assessment of At Risk Mental State (CAARMS) | "Month1"
  A tool developed by Mc Gorry in 2005 to identify subjects at high risk of developing psychosis, track the evolution of their symptoms and set a symptomatic threshold for the actual transition to psychosis. It is recommended that its administration be reserved for "help seeking" subjects (Schultze-Lutter et al, 2015) and is accompanied by an overall operating quotation by SOFAS. It is divided into 7 scales, and makes it possible to identify 3 phenotypes of UHR subjects: vulnerable group
Comprehensive Assessment of At Risk Mental State (CAARMS) | "Month 12"
  A tool developed by Mc Gorry in 2005 to identify subjects at high risk of developing psychosis, track the evolution of their symptoms and set a symptomatic threshold for the actual transition to psychosis. It is recommended that its administration be reserved for "help seeking" subjects (Schultze-Lutter et al, 2015) and is accompanied by an overall operating quotation by SOFAS. It is divided into 7 scales, and makes it possible to identify 3 phenotypes of UHR subjects: vulnerable group

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Relais Collégiens-Lycéens, La Courneuve
  - URC Ville Evrard, Neuilly-sur-Marne
  - CASADO, Saint-Denis
  - CMP Adulte Saint-Denis, Saint-Denis
  - CMP Adulte Saint-Ouen, Saint-Ouen

IPD SHARING:
Plan to Share IPD: No